CLINICAL TRIAL: NCT01480596
Title: A Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacodynamics of Belimumab in Subjects With Generalized Myasthenia Gravis (MG)
Brief Title: The Evaluation of Belimumab in Myasthenia Gravis (MG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115123
Record Dates: First submitted 2011-10-27; First posted 2011-11-29 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Myasthaenia Gravis
MeSH Terms: interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belimumab (Experimental): 10mg/kg
  Interventions: Biological: Belimumab
- Placebo (Placebo Comparator): placebo IV infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Belimumab — 10mg/kg IV infusion
  Arms: Belimumab
Other: Placebo — placebo IV infusion
  Arms: Placebo

SUMMARY:
Study BEL115123 is a randomized, placebo-controlled, double-blind, multinational study of belimumab (10 mg/kg) to investigate the efficacy and safety of belimumab in subjects with MG. The study will enroll male and female outpatients (> or equal to 18 years of age) with a diagnosis of MG who are 1) acetylcholine receptor (AChR) antibody positive or muscle specific kinase (MuSK) antibody positive, 2) on current standard of care therapy, and 3) continue to exhibit signs of MG. The study will include 3 phases: a 4 week screening period, a 24 week treatment period, and a 12 week follow-up period. IP will be administered intravenously on Days 0, 14, 28 and then every 28 days through and including Week 20. At Week 24, primary outcomes will be obtained. Follow up evaluations will be conducted at Weeks 28, 32 and 36 for all subjects. The primary objective of this study is to assess the efficacy of belimumab as evaluated by the change in the quantitative myasthenia gravis (QMG) score.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, with life expectancy of greater than 1 year.
* MG of class II to IVa inclusive.
* Acetylcholine receptor (AChR) or muscle specific kinase (MuSK) antibody positive.
* Stable dose (defined as no dose changes) not exceeding the maximum doses given in Section 5.6.1 of the following therapy(ies) prior to screening: Cholinesterase inhibitor(pyridostigmine or equivalent) for at least 2 weeks prior to screening and no immunosuppressants; Cholinesterase inhibitor (pyridostigmine or equivalent) for at least 2 weeks prior to screening and/or only one of the following: prednisone (up to 40 mg/day or equivalent) for at least 1 month prior to screening; azathioprine for at least 6 months prior to screening; mycophenolate for at least 6 months prior to screening, or cyclosporine for at least 3 months prior to screening; or Cholinesterase inhibitor (pyridostigmine or equivalent) for at least 2 weeks prior to screening and/or prednisone (up to 20 mg/day or equivalent) for at least 1 month prior to screening and only one of the following: azathioprine for at least 6 months prior to screening, mycophenolate for at least 6 months prior to screening, or cyclosporine for at least 3 months prior to screening
* Quantitative Myasthenia Gravis (QMG) score of 8 or greater, with at least 4 points derived from signs other than ocular
* A female subject is eligible to participate if she is: Of non-childbearing potential; Of childbearing potential and NOT pregnant or nursing, has a negative serum pregnancy test at screening, and agrees to one of the following: Complete abstinence from penile-vaginal intercourse, when this is the female's preferred and usual lifestyle, for the period from consent into the study until 16 weeks after the last dose of investigational product; or Consistent and correct use of one of the following acceptable methods of birth control for the period from consent into the study until 16 weeks after the last dose of investigational product: Oral contraceptives (either combined or progesterone only), Injectable progesterone, Implants of etonogestrel or levonorgestrel, Estrogenic vaginal ring, Percutaneous contraceptive patches, Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year, Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study; this male must be the sole partner for the subject, Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Single QTc less than 450 msec; or QTc less than 480 msec in subjects with Bundle Branch Block.
* AST and ALT less than 2xULN; alkaline phosphatase and bilirubin less or = to 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).

Exclusion Criteria:

* Participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) prior to screening or planning to take any investigational drug for the planned duration of study participation (6 months after the last dose of study drug).
* Presence or previous history of thymoma.
* Thymectomy within 12 months
* Clinically significant (in the opinion of investigator) abnormal laboratory values.
* Pregnant females as determined by positive (serum) hCG test at screening or prior to dosing, or lactating females or planning to become pregnant within 16 weeks after last dose of investigational product.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* May require (in the opinion of investigator) treatment with IVIg and/or plasmapheresis during the 24 week treatment period.
* Have received IVIg and/or plasmapheresis within 90 days prior to screening.
* Have received any other biopharmaceutical agent (except IVIg as described in exclusion criteria #8) in the 364 days prior to screening.
* Have received treatment with any B cell targeted therapy (e.g., rituximab, belimumab), at any time.
* Have received a live vaccine within 30 days of study Day 0 (baseline).
* Have received cyclophosphamide or any other immunosuppressive agent apart from the ones allowed by the inclusion criteria #4, within the past 6 months.
* Have another medical condition that requires treatment with steroids or immunosuppressive agents.
* Hospitalization due to infection or use of parenteral antibacterial, antifungal or antiviral agents within 60 days prior to screening; or history of recurrent or chronic infection, or currently active systemic infection.
* Have a history of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Have a history of a major organ transplant (eg, heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Have a historically positive test or test positive at screening for HIV-1, hepatitis B surface antigen or hepatitis C antibody.
* Have an IgG Grade 3 or greater deficiency (less than or = to 400mg/dL).
* Have an IgA deficiency (IgA less than 10mg/dL).
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
* Has a progressive medical, neurological or psychological condition or situation that, in the investigator's judgment, is likely to cause the subject to be unable or unwilling to participate in study procedures, to complete all scheduled assessments, or precludes accurate assessments.
* Is currently abusing drugs or alcohol or has history of abuse in the last 12 months.
* Subjects who have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation of type 4 or 5 on the C-SSRS in the last 2 months or who in the investigator's judgment, pose a significant suicide risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- United States (15):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Burlington, Vermont
  - GSK Investigational Site, Charlottesville, Virginia
- Canada (4):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
- Germany (4):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- Italy (2):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy

REFERENCES:
- [Derived] Hewett K, Sanders DB, Grove RA, Broderick CL, Rudo TJ, Bassiri A, Zvartau-Hind M, Bril V; BEL115123 Study Group. Randomized study of adjunctive belimumab in participants with generalized myasthenia gravis. Neurology. 2018 Apr 17;90(16):e1425-e1434. doi: 10.1212/WNL.0000000000005323. Epub 2018 Mar 21. PMID 29661905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) with myasthenia gravis (MG) and who were acetylcholine receptor (AChR) or muscle-specific kinase (MuSK) antibody positive, on current standard of care therapy and continued to exhibit signs of MG were eligible for participation in the study.
Pre-assignment Details: The study was conducted in 3 phases: a 4 week screening period, a 24 week Treatment (trt) Period, and a 12 week Follow-up period. A total of 40 par. were enrolled, however 1 par. withdrew due to MG exacerbation on Day 7 prior to the first efficacy assessment; therefore, 39 par. comprise the Intent-to-Treat (ITT) Population.
Groups:
- Placebo IV: Participants received 250 milliliter (ml) of a normal saline placebo administered as intravenous (IV) infusion on Days 0, 14, 28 and then every 28 days through Week 20 of the treatment period. Participants continued with the standard of care therapy throughout the treatment period.
- Belimumab 10 mg/kg IV: Participants received 10 milligrams per kilogram (mg/kg) of belimumab administered as IV infusion in 250 mL normal saline on Days 0, 14, 28 and then every 28 days through Week 20 of the treatment period. Participants continued with the standard of care therapy throughout the treatment period.
Period: Overall Study
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Started | 22 | 18
Completed | 17 | 16
Not Completed | 5 | 2
Not completed — Adverse Event | 3 | 0
Not completed — MG exacerbation or change in medication | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo IV: Participants received 250 ml of a normal saline placebo administered as IV infusion on Days 0, 14, 28 and then every 28 days through Week 20 of the treatment period. Participants continued with the standard of care therapy throughout the treatment period.
- Belimumab 10 mg/kg IV: Participants received 10 mg/kg of belimumab administered as IV infusion in 250 mL normal saline on Days 0, 14, 28 and then every 28 days through Week 20 of the treatment period. Participants continued with the standard of care therapy throughout the treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.0 (13.88) | 52.7 (17.32) | 56.1 (15.67)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 7 | 8 | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian - East Asian Heritage | 1 | 1 | 2
  White - White/Caucasian/European Heritage | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline for Quantitative Myasthenia Gravis (QMG) Score at Week 24
Description: The QMG is a 13 item ordinal scale which measures ocular, bulbar, extremity fatigue and strength, along with respiratory function. The total QMG score was calculated by adding the score of each of the 13 individual QMG questions. Possible scoring on the QMG range from 0 (normal) to 39 (severe). A lower score indicates a better clinical outcome. The QMG score at Baseline is the average of the screening and Week 0 Baseline scores. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. The differences in adjusted least square means were presented (Belimumab 10 mg/kg minus Placebo). A negative treatment difference indicates benefit relative to placebo. The analysis method was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline QMG Score, Treatment by Visit, and Baseline QMG Score by Visit.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population includes participants in the Safety Population who has provided any post treatment efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 17 | 17
Units on a scale | -2.37 (1.099) | -4.21 (1.143)
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.256, Mixed Models Analysis; Mean Difference (Final Values) = -1.84, 95% CI 2-sided [-5.08 to 1.40], Standard Error of Mean 1.592 — Standard error of mean is for adjusted difference

2. Secondary Outcome: Number of Participants With Improvement by Greater Than or Equal to (>=) 3 Points From Baseline Through to Week 24 in the QMG Score
Description: The QMG is a 13 item ordinal scale which measures ocular, bulbar, extremity fatigue and strength, along with respiratory function. The total QMG score was calculated by adding the score of each of the 13 individual QMG questions. Possible scoring on the QMG range from 0 (normal) to 39 (severe). A lower score indicates a better clinical outcome. The QMG score at Baseline is the average of the screening and Week 0 Baseline scores. Proportions compared using exact analyses stratified by the observed median Baseline score (less than or equal to [<=] median, greater than [ >] median). Exact odds ratio, double the exact one-sided p-value and exact confidence intervals were presented. Participants with missing data were assumed to have a negative response.
Time Frame: Baseline and up to Week 24
Population: ITT Population.
Measure: Number; unit: Number of participants
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 21 | 18
Number of participants | 6 | 11
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.082, exact methods; Odds Ratio (OR) = 3.81, 95% CI [0.87 to 19.02]

3. Secondary Outcome: Number of Participants Worsening by >=3 Points in QMG Score From Baseline Through to Week 24
Description: The QMG is a 13 item ordinal scale which measures ocular, bulbar, extremity fatigue and strength, along with respiratory function. The total QMG score was calculated by adding the score of each of the 13 individual QMG questions. Possible scoring on the QMG range from 0 (normal) to 39 (severe). A lower score indicates a better clinical outcome. The QMG score at Baseline is the average of the screening and Week 0 Baseline scores. Proportions compared using exact analyses stratified by the observed median Baseline score (<=median, > median). Exact odds ratio, double the exact one-sided p-value and exact confidence interval were presented. Participants with missing data were assumed to have a worsening response.
Time Frame: Baseline and up to Week 24
Population: ITT Population.
Measure: Number; unit: Number of participants
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 21 | 18
Number of participants | 4 | 2
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.827, exact methods; Odds Ratio (OR) = 0.55, 95% CI [0.05 to 4.35]

4. Secondary Outcome: Number of Participants With a Sustained Response in the QMG Score
Description: A sustained response during the treatment phase is when a participant improves by >=3 points from Baseline at Week 12, and the participant maintains at least a 3 point improvement from Baseline through Week 24. The QMG is a 13 item ordinal scale which measures ocular, bulbar, extremity fatigue and strength, along with respiratory function. The total QMG score was calculated by adding the score of each of the 13 individual QMG questions. Possible scoring on the QMG range from 0 (normal) to 39 (severe). A lower score indicates a better clinical outcome. The QMG score at Baseline is the average of the screening and Week 0 Baseline scores. Odds ratios are calculated by Cochran-Mantel-Haenszel method stratified by the observed median baseline score (<= median, > median). Wald confidence intervals and p-values were presented.
Time Frame: Baseline and up to Week 24
Population: ITT Population.
Measure: Number; unit: Number of participants
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 21 | 18
Number of participants | 5 | 8
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.184, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.51, 95% CI 2-sided [0.62 to 10.10]

5. Secondary Outcome: Median Time to QMG Response Which is Sustained From Earliest Time Point at Which Improvement by >=3 Points From Baseline is Observed and Maintained Through Week 24
Description: A sustained response during the treatment phase is when a participant improves by >=3 points from Baseline at Week 12, and the participant maintains at least a 3 point improvement from Baseline through Week 24. The QMG is a 13 item ordinal scale which measures ocular, bulbar, extremity fatigue and strength, along with respiratory function. The total QMG score was calculated by adding the score of each of the 13 individual QMG questions. Possible scoring on the QMG range from 0 (normal) to 39 (severe). A lower score indicates a better clinical outcome. The QMG score at Baseline is the average of the screening and Week 0 Baseline scores.
Time Frame: Baseline and up to Week 24
Population: As per the criteria documented in the Reporting and Analysis Plan these analyses were not conducted since <50% of subjects met the criteria (i.e. had the event in question).
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mean Change From Baseline for QMG Score at Week 28, Week 32 and Week 36
Description: The QMG is a 13 item ordinal scale which measures ocular, bulbar, extremity fatigue and strength, along with respiratory function. Total QMG score was calculated by adding the score of each of the 13 individual QMG questions. Possible scoring on the QMG range from 0 (mild) to 39 (severe). A lower score indicates a better clinical outcome. The QMG score at baseline (BL) is the average of the screening and Week 0 BL scores. Change from BL was calculated by subtracting the BL value from the post-BL value. The differences in adjusted least square means are presented (Belimumab 10 mg/kg minus Placebo). A negative trt difference indicates benefit relative to placebo. Analysis method was Mixed-Model Repeated Measures adjusted for Trt, Visit, BL QMG Score, Trt by Visit and BL QMG Score by Visit. Only follow-up visits are presented but the analysis also includes all trt phase visits. Only those par. available at indicated time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline, Week 28, Week 32 and Week 36
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 21 | 18
Units on a scale
  Week 28, n=16, 14 | -3.33 (0.839) | -5.03 (0.889)
  Week 32, n=15, 16 | -2.82 (0.880) | -4.12 (0.904)
  Week 36, n=17, 14 | -2.44 (0.872) | -4.73 (0.921)
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.175, Mixed Models Analysis; Mean Difference (Final Values) = -1.70, 95% CI 2-sided [-4.20 to 0.80], Standard Error of Mean 1.228 — Analysis for Week 28. Standard error of mean is for adjusted difference
Statistical Analysis 2: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.310, Mixed Models Analysis; Median Difference (Final Values) = -1.31, 95% CI 2-sided [-3.89 to 1.28], Standard Error of Mean 1.267 — Analysis for Week 32. Standard error of mean is for adjusted difference
Statistical Analysis 3: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis; Median Difference (Final Values) = -2.29, 95% CI 2-sided [-4.88 to 0.30], Standard Error of Mean 1.272 — Analysis for Week 36. Standard error of mean is for adjusted difference

7. Secondary Outcome: Mean Change From Baseline in Myasthenia Gravis Composite (MGC) Scale Through to Week 24
Description: The total MGC score was calculated by adding the score of each of the 10 individual MGC questions. Possible total MGC scores range from 0 (normal) to 50 (severe). A lower score indicates a better clinical outcome. Baseline is defined as the participants last available assessment prior to initiation of study IV infusion. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. The differences in adjusted least square means are presented (Belimumab 10 mg/kg minus Placebo). A negative treatment difference indicates benefit relative to placebo. The analysis method was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline MGC Score, Treatment by Visit, and Baseline MGC Score by Visit.
Time Frame: Baseline and up to Week 24
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 17 | 17
Units on a scale | -3.86 (1.037) | -3.81 (1.064)
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.972, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-2.97 to 3.07], Standard Error of Mean 1.486 — Standard error of mean is for adjusted difference

8. Secondary Outcome: Number of Participants With Improvement by >=3 Points From Baseline Through to Week 24 in the MGC Score
Description: The total MGC score was calculated by adding the score of each of the 10 individual MGC questions. Possible total MGC scores range from 0 (normal) to 50 (severe). A lower score indicates a better clinical outcome. Baseline is defined as the participants last available assessment prior to initiation of study IV infusion. Proportions compared using exact analyses stratified by the observed median baseline score (<= median, > median). Exact odds ratios, double the exact one-sided p-values and exact confidence intervals were presented. Participants with missing data were assumed to have a negative response.
Time Frame: Baseline and up to Week 24
Population: ITT Population.
Measure: Number; unit: Number of participants
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 21 | 18
Number of participants | 10 | 9
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 1.000, exact methods; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.26 to 5.48]

9. Secondary Outcome: Number of Participants Worsening by >=3 Points From Baseline Through to Week 24 in the MGC Score
Description: The total MGC score was calculated by adding the score of each of the 10 individual MGC questions. Possible total MGC scores range from 0 (normal) to 50 (severe). A lower score indicates a better clinical outcome. Baseline is defined as the participants last available assessment prior to initiation of study IV infusion. Proportions compared using exact analyses stratified by the observed median baseline score (<= median, > median). Exact odds ratios, double the exact one-sided p-values and exact confidence intervals were presented. Participants with missing data were assumed to have a worsening response.
Time Frame: Baseline and up to Week 24
Population: ITT Population.
Measure: Number; unit: Number of participants
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 21 | 18
Number of participants | 5 | 2
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.530, exact methods; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.03 to 2.89]

10. Secondary Outcome: Number of Participants With a Sustained Response in the MGC Score
Description: AA sustained response during the treatment phase is when a participant improves by >=3 points from Baseline at Week 12, and the participant maintains at least a 3 point improvement from Baseline through Week 24. The total MGC score was calculated by adding the score of each of the 10 individual MGC questions. Possible total MGC scores range from 0 (normal) to 50 (severe). A lower score indicates a better clinical outcome. Baseline is defined as the participants last available assessment prior to initiation of study IV infusion. Odds ratios are calculated by Cochran-Mantel-Haenszel method without adjusting for any strata. Wald confidence intervals and p-values were presented.
Time Frame: Baseline and up to Week 24
Population: ITT Population.
Measure: Number; unit: Number of participants
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 21 | 18
Number of participants | 4 | 7
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.175, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.70, 95% CI 2-sided [0.64 to 11.46]

11. Secondary Outcome: Median Time to MGC Response Which is Sustained From Earliest Time Point at Which Improvement by >=3 Points From Baseline is Observed and Maintained Through Week 24
Description: A sustained response during the treatment phase is when a participant improves by >=3 points from Baseline at Week 12, and the participant maintains at least a 3 point improvement from Baseline through Week 24. The total MGC score was calculated by adding the score of each of the 10 individual MGC questions. Possible total MGC scores range from 0 (normal) to 50 (severe). A lower score indicates a better clinical outcome. Baseline is defined as the participants' last available assessment prior to initiation of study intravenous (IV) infusion.
Time Frame: Baseline and up to Week 24
Population: as for outcome 5
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Mean Change From Baseline for MGC Score at Week 28, Week 32 and Week 36
Description: The total MGC score was calculated by adding the score of each of the 10 individual MGC questions. Possible total MGC scores range from 0 (normal) to 50 (severe). A lower score indicates a better clinical outcome. Baseline is defined as the participant's last available assessment prior to initiation of study IV infusion. Change from Baseline was calculated by subtracting the Baseline value from the post-BL value. The differences in adjusted least square means are presented (Belimumab 10 mg/kg minus Placebo). A negative treatment difference indicates benefit relative to placebo. The analysis method was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline MGC Score, Treatment by Visit, and Baseline MGC Score by Visit. Only follow-up visits are presented but the analysis also includes all treatment phase visits. Only those participants available at the indicated time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline, Week 28, Week 32 and Week 36
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 21 | 18
Units on a scale
  Week 28, n=16, 14 | -4.63 (0.856) | -5.64 (0.905)
  Week 32, n=15, 16 | -5.46 (0.975) | -5.44 (0.948)
  Week 36, n=17, 14 | -4.77 (0.970) | -5.04 (1.052)
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.423, Mixed Models Analysis; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-3.56 to 1.53], Standard Error of Mean 1.245 — Analysis for Week 28. Standard error of mean is for adjusted difference
Statistical Analysis 2: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.986, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-2.76 to 2.80], Standard Error of Mean 1.361 — Analysis for Week 32. Standard error of mean is for adjusted difference
Statistical Analysis 3: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.848, Mixed Models Analysis; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-3.21 to 2.65], Standard Error of Mean 1.430 — Analysis for Week 36. Standard error of mean is for adjusted difference

13. Secondary Outcome: Number of Participants With a Myasthenia Foundation of America-post Intervention Status (MGFA-PIS) of Minimal Manifestation or Better at Week 24 and Week 36.
Description: Myasthenia Foundation of America-post intervention status assesses whether subjects can be categorized as being in a status of Minimal Manifestation (MM), Pharmacologic Remission (PR) or Complete Remission (CR). Only MM and PR were assessed in this study as CR is not achievable based on the definition.
Time Frame: Week 24 and Week 36
Population: The Reporting and Analysis Plan pre-specified that these analyses would not be conducted since during a review of blinded data it was identified that the MGFA scale had been inconsistently performed across sites and any statistical analyses would not be interpretable.
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Participants With MGFA-PIS of Pharmacologic Remission or Better at Week 24 and Week 36
Description: Myasthenia Foundation of America (MGFA) post intervention status (PIS) assesses whether subjects can be categorized as being in a status of Minimal Manifestation (MM), Pharmacologic Remission (PR) or Complete Remission (CR). Only MM and PR were assessed in this study as CR is not achievable based on the definition.
Time Frame: Week 24 and Week 36
Population: as for outcome 13
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With MGFA-PIS of Minimal Manifestation Sustained Response (MM at Week 12 and Maintained the Response Through Week 24)
Description: as for outcome 14
Time Frame: Week 12 through Week 24
Population: as for outcome 13
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Number of Participants With MGFA-PIS of Pharmacologic Response Sustained Response (PR at Week 12 and Maintained the Response Through Week 24)
Description: as for outcome 14
Time Frame: Week 12 through Week 24
Population: as for outcome 13
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Participants With MGFA-PIS (Unchanged, Improved, Worsened) at Week 24 and Week 36
Description: Myasthenia Foundation of America (MGFA) post intervention status (PIS) assesses whether subjects can be categorized as being unchanged, improved or worsened.
Time Frame: Week 24 and Week 36
Population: as for outcome 13
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Mean Change From Baseline in the Myasthenia Gravis Activities of Daily Living Scale (MG-ADL) at Week 12 and Week 24
Description: The total MG-ADL score was calculated by adding the score of each of the 8 individual MG-ADL questions. Possible total MG-ADL scores ranges from 0 (normal) to 24 (severe). A lower score indicates a better clinical outcome. Baseline is defined as the participants last available assessment prior to initiation of study IV infusion. Change from Baseline was calculated by subtracting the Baseline value from the post-baseline value. The differences in adjusted least square means are presented (Belimumab 10 mg/kg minus Placebo). A negative treatment difference indicates benefit relative to placebo. The analysis method was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline MG-ADL Score, Treatment by Visit, and Baseline MG-ADL Score by Visit. Only those participants available at the indicated time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 21 | 18
Units on a scale
  Week 12, n=19, 18 | -1.33 (0.489) | -1.83 (0.511)
  Week 24, n=17, 17 | -2.01 (0.589) | -2.32 (0.603)
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.483, Mixed Models Analysis; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.94 to 0.93], Standard Error of Mean 0.707 — Statistical analysis is presented for Week 12. Standard error of mean is for adjusted mean difference
Statistical Analysis 2: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.711, Mixed Models Analysis; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-2.03 to 1.40], Standard Error of Mean 0.844 — Statistical analysis is presented for Week 24. Standard error of mean is for adjusted mean difference

19. Secondary Outcome: Mean Change From Baseline in the Myasthenia Gravis Activities of Daily Living Scale (MG-ADL) at Week 28, Week 32 and Week 36
Description: The total MG-ADL score was calculated by adding the score of each of the 8 individual MG-ADL questions. Possible total MG-ADL scores range from 0 (normal) to 24 (severe). A lower score indicates a better clinical outcome. Baseline is defined as the participant's last available assessment prior to initiation of study IV infusion. Change from Baseline was calculated by subtracting the Baseline value from the post-Baseline value. The differences in adjusted least square means are presented (Belimumab 10 mg/kg minus Placebo). A negative treatment difference indicates benefit relative to placebo. The analysis method was Mixed-Model Repeated Measures adjusted for Treatment, Visit, Baseline MG-ADL Score, Treatment by Visit, and Baseline MG-ADL Score by Visit. Only follow-up visits are presented but the analysis also includes all treatment phase visits. Only those participants available at the indicated time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline, Week 28, Week 32 and Week 36
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Number analyzed (Participants) | 21 | 18
Units on a scale
  Week 28, n=16, 14 | -1.21 (0.522) | -2.96 (0.546)
  Week 32, n=15, 16 | -1.52 (0.632) | -1.80 (0.619)
  Week 36, n=17, 14 | -1.51 (0.621) | -1.78 (0.663)
Statistical Analysis 1: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.028, Mixed Models Analysis; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-3.30 to -0.20], Standard Error of Mean 0.757 — Analysis for Week 28. Standard error of mean is for adjusted difference
Statistical Analysis 2: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.756, Mixed Models Analysis; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-2.10 to 1.55], Standard Error of Mean 0.887 — Analysis for Week 32. Standard error of mean is for adjusted difference
Statistical Analysis 3: Comparison: Placebo IV vs Belimumab 10 mg/kg IV; Test type: Superiority or Other; p = 0.775, Mixed Models Analysis; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-2.12 to 1.59], Standard Error of Mean 0.909 — Analysis for Week 36. Standard error of mean is for adjusted difference

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs were collected from the date first infusion of investigational product up to the Week 24 visit.
Description: AEs and SAEs are reported for the safety population which is comprised of participants who had at least one infusion of study agent.
Arm/Group | Placebo IV | Belimumab 10 mg/kg IV
Serious Adverse Events (participants affected / at risk) | 4/22 | 0/18
Other Adverse Events (participants affected / at risk) | 16/22 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo IV (N=22) | Belimumab 10 mg/kg IV (N=18)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Aortic dissection rupture (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo IV (N=22) | Belimumab 10 mg/kg IV (N=18)
Influenza (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Cystitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 2
Fatigue (General disorders) | 0 | 1
Feeling hot (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Eye pain (Eye disorders) | 0 | 1
Photopsia (Eye disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Neutrophil count increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.